CLINICAL TRIAL: NCT01631903
Title: A Phase 2, Multi-Center, Five-Arm, Parallel Design, Randomized, Single-Blind Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Proellex® (Telapristone Acetate) Administered Vaginally in the Treatment of Premenopausal Women With Uterine Fibroids Confirmed by Ultrasound
Brief Title: Extension of Study ZPV-200
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ZPV-200 EXT
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2012-11

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — telapristone acetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 2 (3mg) (Experimental)
  Interventions: Drug: telepristone acetate 3 mg
- Arm 3 (6 mg) (Experimental)
  Interventions: Drug: telepristone acetate 6 mg
- Arm 4 (12 mg) (Experimental)
  Interventions: Drug: telepristone acetate 12 mg
- Arm 5 (24 mg) (Experimental)
  Interventions: Drug: telepristone acetate 24 mg
- PK arm (12 mg) (Experimental): PK arm requires one additional 24 hour PK assessment at V3 and daily visits between visits 2 and 3 for drug trough sample collection
  Interventions: Drug: telepristone acetate 12 mg

INTERVENTIONS:
Drug: telepristone acetate 12 mg — 12 mg, vaginal capsule, once daily for 4 months
  Other Names: Proellex
  Arms: PK arm (12 mg)
Drug: telepristone acetate 3 mg — 3 mg, vaginal capsule, once daily for 3 months
  Other Names: Proellex
  Arms: Arm 2 (3mg)
Drug: telepristone acetate 6 mg — 6 mg, vaginal capsule, once daily for 3 months
  Other Names: Proellex
  Arms: Arm 3 (6 mg)
Drug: telepristone acetate 12 mg — 12 mg, vaginal capsule, once daily, for 3 months
  Other Names: Proellex
  Arms: Arm 4 (12 mg)
Drug: telepristone acetate 24 mg — 24 mg, vaginal capsule, once daily for 4 months
  Other Names: Proellex
  Arms: Arm 5 (24 mg)

SUMMARY:
The purpose of this study is to determine the safety, pharmacokinetics and efficacy of four doses of vaginally administered Proellex in premenopausal women with uterine fibroids confirmed by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult females between 18 and 47 years of age with uterine fibroids confirmed by ultrasound. Normal, or abnormal but non-clinically significant, transvaginal ultrasound. History of menstrual events occurring in regular cycles.
* Agreement not to attempt to become pregnant.
* Agreement to limit alcohol consumption to no more than 2 drinks per week and to avoid alcohol consumption within 48 hours before each visit.
* Ability to complete a daily subject diary and study procedures in compliance with the protocol.
* Agrees to use the condoms provided and no other method of birth control (hormonal methods, contraceptive sponge, spermicide or cervical cap) over the course of the study.
* Has a negative pregnancy test at the Screening and Baseline visits. An exception for the pregnancy test requirement will be granted for subjects providing verification of surgical sterilization.
* A Body Mass Index (BMI) between 18 and 39 inclusive.
* Is available for all treatment and follow-up visits.
* Subject is able to insert vaginal suppositories.
* Subject is willing to exclusively use sanitary napkins (no tampons) during study duration.

Exclusion Criteria:

* Subject is a post-menopausal woman, defined as either; six (6) months or more (immediately prior to screening visit) without a menstrual period, or prior hysterectomy and/or oophorectomy.
* Subject is pregnant or lactating or is attempting or expecting to become pregnant during the 7 month study period.
* Women with abnormally high liver enzymes or liver disease. (ALT or AST exceeding 1.5x ULN AND total bilirubin exceeding 1.5xULN at screening and confirmed on repeat).
* Received an investigational drug in the 30 days prior to the screening for this study.
* Women with a history of PCOS.
* Concurrent use of any testosterone, progestin, androgen, estrogen, anabolic steroids, DHEA or hormonal products for at least 2 weeks prior to screening and during the study.
* Use of oral contraceptives in the preceding 30 days. Use of Depo-Provera® in the preceding 6 months.
* Has an IUD in place.
* Women currently using narcotics.
* Women currently taking cimetidine or spironolactone.
* Clinically significant abnormal findings on screening examination or any condition, which in the opinion of the investigator, would interfere with the participant's ability to comply with the study instructions or endanger the participant if she took part in the study.
* Participation in study ZP-204.

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Bleeding Scores | 3 or 4 months depending on treatment arm
  The primary efficacy endpoint will be bleeding assessed using the change in PBAC scores from the 4 weeks prior to Visit 2 to the 4 weeks prior to Visit 10

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Miami Gardens, Florida
  - Houston, Texas

REFERENCES:
- See also: Sponsor's corporate web page — http://www.reprosrx.com